CLINICAL TRIAL: NCT06803667
Title: Use of the Moving Shot Radiofrequency Ablation Technique for the Treatment of Vascular Anomalies
Brief Title: Radiofrequency Ablation of Vascular Anomalies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Edward Gayou, Edward Gayou MD, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-55373
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Vascular Anomalies
Keywords: Venous Malformation; Lymphatic Malformation; Vascular Anomaly; Radiofrequency Ablation
MeSH Terms: conditions — Vascular Malformations; Lymphatic Abnormalities | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiofrequency Ablation Treatment (Experimental): Participants in this single arm study will undergo percutaneous radiofrequency ablation of their vascular anomaly.
  Interventions: Device: Radiofrequency ablation alone

INTERVENTIONS:
Device: Radiofrequency ablation alone — Radiofrequency ablation under imaging guidance allows for heating of diseased tissues, and has been used for the treatment of benign and malignant soft tissue masses throughout the body in the United States over the last several decades. Newer radiofrequency ablation devices are smaller and allow for precision temperature regulation; these technologies allow us to safely and precisely deliver heat to diseased tissues while minimizing the heating of nearby healthy tissues. Furthermore, we are able to clearly see these devices under ultrasound, which allows us to move the device in real-time to deliver heat as safely, effectively, and efficiently as possible.

SUMMARY:
Vascular Anomalies (VA) are areas of disorganized blood vessel tissue that can appear as lumps or bumps under the skin. Sometimes they can cause you discomfort, or you may not like how they look. One option for treatment is to place a needle through the skin into the VA and inject medicines called sclerosants that can cause them to shrink. This treatment is called sclerotherapy and is the standard of care. While sclerotherapy is safe and effective, other alternatives for treatment exist, such as using heat. Just like with sclerotherapy, a small needle is inserted through the skin into the VA while the doctor watches it using imaging techniques. Once the needle tip is in the right spot, the needle tip delivers heat energy to the VA, causing it to shrink. We believe that using heat to treat VAs may be safer and more effective than using sclerotherapy, and we are asking for your participation in this study to help us determine whether that is correct.

You are being given the option of using heat instead of sclerosant medicines to treat your VA. Regardless of whether you choose targeted heat or sclerosant medicine injection for your treatment, all procedures will be performed under sedation with an anesthesiologist, and you will continue to have appointments with the vascular anomalies clinic after your procedure.

The risks to you if you decide to use heat for treatment of your vascular anomaly are similar to injecting sclerosant medicines, which includes bleeding, infection, and damage to nearby structures.

There is also the additional risk of heating the skin and causing a burn, but the risk of this is low.

Benefits of using heat instead of sclerosant medicine include avoiding sclerosant medicine side effects. Possible benefits include more effective treatment of your vascular anomaly than could be achieved with traditional sclerotherapy.

Participation is entirely voluntary, and if you decide not to use heat for treatment of your VA, you are free to discuss with your doctor alternative treatments like sclerotherapy.

DETAILED DESCRIPTION:
Patients who seek care for their vascular anomalies at the Texas Children's Vascular Anomalies (VA) clinic will be potentially eligible for this study. Patients who are diagnosed with a VA and interested in having it treated will be discussed among the vascular anomalies clinic physicians. If vascular anomalies clinic physicians feel that heating the vascular anomaly using a radiofrequency needle is a good option, you will then be offered heat ablation as an alternative to sclerotherapy. After a risks and benefits discussion, if you are interested in having your vascular anomaly treated with heat instead of sclerotherapy, you will be enrolled. You will be asked to rate your pain on a scale of 1-10 when your pain is at its worst, 1 being no pain at all, and 10 being the worst pain imaginable.

Once enrolled, you will be scheduled for your procedure date. Procedures are typically scheduled in the morning, and you will be asked to fast after midnight. When you arrive for your procedure, you will be evaluated by the anesthesia team, and an appropriate sedation plan will be determined. Once all safety checks are performed, you will be taken back into one of the interventional radiology suites, and you will receive anesthesia medicine. Once the medicine has been administered, you will be positioned on the interventional radiology table. A plastic pad will be carefully placed on each of your thighs. These are called grounding pads and allow for the radiofrequency ablation probe to generate heat energy when activated.

Once the pads are safely secured on the thighs, your skin directly above the vascular anomaly will be prepped with cleaning solution, and sterile drapes will be placed to reduce the risk of infection. Once the final safety check is performed, the procedure will begin. Using a special imaging tool called ultrasound that uses sound waves to allow us to see structures under the skin, the operator will identify the vascular anomaly. Then, while watching under ultrasound, the ablation needle will carefully be inserted into the vascular anomaly. Once the operator is satisfied with the position of the radiofrequency ablation needle, the device will be turned on, and heat will be delivered to the vascular anomaly. The needle will be moved slightly to ensure that heat reaches all parts of the vascular anomaly. We always watch the ablation needle whenever it is actively delivering heat or when we are moving it to reduce the risk of heating other areas near the vascular anomaly. Once the vascular anomaly has been sufficiently heated, the needle will be removed, and a small bandage will be placed. You will then be taken to the recovery area, where you will be allowed to go home after the effects of the anesthesia have ended.

You will meet with the physician who performed the procedure 1 week postoperatively for a virtual clinic visit for a check-in. If all is well at this virtual clinic appointment, you will then return in person 8 weeks after your treatment date. During this clinic visit, you will be evaluated by vascular anomalies clinic physicians, and you will be asked to rate your pain on a scale of 1-10, as described earlier. In addition to that, you will have an ultrasound performed on the vascular anomaly, so we can assess the effects of the heat and compare it to before the procedure. You will have another in person vascular anomalies clinic at 6 months following the treatment date, which will be identical to the 2 month clinic visit. After this 6 month clinic visit, your participation will be concluded. In total, we expect your participation in this study to last about 6 months, measured from enrollment after first clinic visit, to the 3rd and final 6 month postoperative clinic visit. However, it may be slightly longer than this depending on the scheduling of the ablation procedure and subsequent clinic visits. Participation in this trial is entirely voluntary, you may choose to stop participating at any time.

ELIGIBILITY:
Inclusion Criteria

Patients Over Three Years of Age

Radiologic Diagnosis of "Slow Flow" Vascular Malformation, using either Doppler Ultrasound and/or MRI, that is a candidate for sclerotherapy treatment after discussion in multidisciplinary committee

Vascular Malformations are a subset of Vascular Anomalies as defined by the International Society For the Study of Vascular Anomalies of 2018 Classification

Vascular Malformations Include:

Capillary Malformations Lymphatic Malformations Venous Malformations Arteriovenous Malformations Arteriovenous Fistula

"Slow Flow" Vascular Malformations, as defined by lack of arterial flow on Duplex Ultrasound, will be eligible for enrollment. These include: Lymphatic Malformations Venous Malformations

Patient is symptomatic (pain, swelling, functionally limited, or cosmetic concern), and Patient/Guardian desires treatment

RFA considered technically feasible and an alternative to targeted sclerotherapy after discussion by multidisciplinary committee

Target "Slow Flow" Vascular Malformation is easily visualized/well characterized with ultrasound such that lesion can be easily targeted for RFA using the "moving shot" technique

Target Area of "Slow Flow" Vascular Malformation is at least 3 mm below the skin surface

Target Area of "Slow Flow" Vascular Malformation is at least 3 mm away from critical neurovascular structures

Patient able to undergo General Anesthesia

Patient/Guardian Agreeable to RFA in lieu of percutaneous sclerotherapy

Patients who have had their vascular anomalies previously treated as well as treatment naive patients are all eligible.

Exclusion Criteria

History of metallic surgical implants (Pacemaker, ICD, Implantable pain Pump, Spinal cord Stimulator ETC)

Pregnant Patients All patients who have begun their menstrual cycle OR are 12 years of age or older will be asked to perform a pregnancy test, either urine or blood per our institutional protocols. If patient/family refuses, signed acknowledgement will be obtained that documents refusal and affirmation of non-pregnant status

Patient unable to safely undergo anesthesia

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pre-procedural ultrasound volume of the lesion of interest, compared with post procedure ultrasound volume of the lesion of interest. | From Enrollment to End of Treament at ~6 Months
  * Pre-procedural ultrasound volume of the lesion of interest, compared with post procedure ultrasound volume of the lesion of interest.
  * This will be measured in cm3 on ultrasound (LxWxHx.05).
  * Pre-procedure will be measured prior to ablation.
  * Post Procedure measurements will occur at 2 month and 6 month postoperative clinic visits.
  * Volume will be summarized and reported in cubic centimeters

SECONDARY OUTCOMES:
Society of Interventional Radiology (SIR) Adverse Event Classification System | Within 30 Days of Procedure Date
  Procedure Related Adverse Events
National Cancer Institute Terminology Criteria for Adverse Events | From Treatment to end of follow-up at ~6 Months

OTHER OUTCOMES:
Visual Analogue Scale Pain Score | Performed prior to procedure and at 2 month and 6 month clinic visits

IPD SHARING:
Plan to Share IPD: Undecided